CLINICAL TRIAL: NCT04573764
Title: Acute Effects of Oral Ketone Ester on Cardiac Function in Patients With COVID-19
Acronym: KetoCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-20021500
Record Dates: First submitted 2020-10-01; First posted 2020-10-05 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — beta-hydroxybutyrate-1,3-butanediol monoester

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blinded crossed-over acute intervention study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-beta-hydroxybutyrate-(R)-1,3 butanediol monoester (Active Comparator)
  Interventions: Dietary Supplement: D-beta-hydroxybutyrate-(R)-1,3 butanediol monoester
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: D-beta-hydroxybutyrate-(R)-1,3 butanediol monoester — The intervention is D-beta-hydroxybutyrate-(R)-1,3 butanediol monoester and will be bought commercially. As an example: One bottle of "KetoneAid KE4 PRO" with 60 ml contains 30 g D-beta-hydroxybutyrate-(R)-1,3 butanediol monoester. For more information please refer to: https://shop.ketoneaid.com/collections/all/products/ke4-pro. Placebo will be a taste-matched water solution provided by the company. The placebo solution and the active solution will be prepared in identic bottles and investigators will be blinded.
  Arms: D-beta-hydroxybutyrate-(R)-1,3 butanediol monoester
Dietary Supplement: Placebo — Taste-matched water
  Arms: Placebo

SUMMARY:
Based on Chinese studies, cardiac injury occurs in 20-30% of hospitalized patients and contributes to 40% of deaths. There are many possible mechanisms of cardiac injury in COVID-19 patients and increased myocardial oxygen demand and decreased myocardial oxygen supply are likely contributors to increased risk of myocardial infarction and heart failure. Interventions reducing the risk of cardiac injury are needed.

Ketone bodies, such as 3-hydroxybutyrate and acetoacetate, can maintain ATP production in the heart and brain during starvation. It has been suggested that ketone bodies are more efficient substrates of energy metabolism than glucose, with a lower oxygen consumption per ATP-molecule produced. In addition, the reduction in hospitalizations due to heart failure observed in type 2 diabetes patients treated with sodium-glucose cotransporter 2 inhibitors, is suggested to be partly attributable to increased levels of 3-hydroxybutyrate. Infusion with 3-hydroxybutyrate reaching a plasma level of approximately 3 mM had acute beneficial hemodynamic effects in patients with heart failure and in healthy controls in a study by Nielsen et al. Improved haemodynamics and reduced systemic oxygen consumption might be of great benefit in patients with COVID-19.

The primary endpoint is left ventricular ejection fraction. Secondary endpoints are conventional echocardiography parameters, peripheral blood oxygen saturation, venous blood oxygen saturation and urine creatinine clearance.

The study population are twelve previously hospitalized patients with COVID-19

The study design is a randomized placebo-controlled double-blinded crossed-over acute intervention study.

ELIGIBILITY:
Inclusion Criteria:

- Patients previously hospitalized at hospitals of greater Copenhagen and the Zealand region with a laboratory confirmed diagnosis of COVID-19 > 18 years of age.

Exclusion Criteria:

* Persons not able to cooperate
* Persons unable to understand and sign "informed consent"
* Diagnosis with chronic obstructive pulmonary disease
* Diagnosis with asthma
* Active treatment with sodium-glucose transporter 2 inhibitors
* eGFR < 15 ml/min/1.73m2
* insulin-dependent diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Left Ventricular ejection fraction | 1 hour
  Echocardiography

SECONDARY OUTCOMES:
Global longitudinal strain | 1 hour
  Echocardiography
Cardiac output | 1 hour
  Echocardiography
Peripheral blood oxygen saturation | 5 minutes
  Pulse oximetry
Venous blood oxygen saturation | 5 minutes
  blood gas analysis
Urine creatinine clearance | 12 hours
  Urine will be collected during the two cross-over sessions and urine creatinine will be measured on these two volumes. Creatinine clearance in ml/min/1.73m2 will then be estimated and compared with plasma creatinine for estimating kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Tor Biering-Sørensen, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Please Select, Denmark

IPD SHARING:
Plan to Share IPD: No